CLINICAL TRIAL: NCT02832635
Title: Effectiveness and Safety of Whole-brain Radiotherapy With/Without TMZ Concurrent Chemotherapy or Avoidance of Hippocampus for Patients of Brain Metastases: a Multi-institutional, Randomized Controlled Clinical Trial
Brief Title: A Clinical Trial on Whole-brain Radiotherapy With Temozolomide Concurrent Chemotherapy or Avoidance of Hippocampus for Patients of Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yun-fei Xia, Director of Department of Radiation Oncology, Principal Investigator, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2016-005-01
Record Dates: First submitted 2016-06-14; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-06

CONDITIONS: Brain Metastasis; Radiation Therapy Complication
Keywords: brain metastasis; whole-brain radiotherapy; TMZ; avoidance of hippocampus
MeSH Terms: conditions — Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- WBRT (Experimental): Patients with brain metastases (>3 lesions) ; Whole-brain radiotherapy without avoidance of hippocampus applied.
  Interventions: Radiation: WBRT without avoidance of hippocampus
- WBRT with avoidance of hippocampus (Experimental): Patients with brain metastases (>3 lesions) ; Whole-brain radiotherapy with avoidance of hippocampus applied.
  Interventions: Radiation: WBRT with avoidance of hippocampus
- WBRT with TMZ (Experimental): Patients with brain metastases (>3 lesions) ; Whole-brain radiotherapy with concurrent TMZ chemotherapy applied.
  Interventions: Drug: TMZ; Radiation: WBRT without avoidance of hippocampus
- WBRT with avoidance of hippocampus and TMZ (Experimental): Patients with brain metastases (>3 lesions) ; Whole-brain radiotherapy with avoidance of hippocampus and concurrent TMZ chemotherapy applied.
  Interventions: Drug: TMZ; Radiation: WBRT with avoidance of hippocampus

INTERVENTIONS:
Drug: TMZ — TMZ 75mg/m2/d from the 1st day to the last day of radiotherapy
  Other Names: temozolomide
  Arms: WBRT with TMZ; WBRT with avoidance of hippocampus and TMZ
Radiation: WBRT with avoidance of hippocampus — Whole brain radiotherapy of 30Gy/10f by IMRT (Intensity Modulation Radiated Therapy), with or without boost. The maximum dose of hippocampus should be no more than 18Gy.
  Arms: WBRT with avoidance of hippocampus; WBRT with avoidance of hippocampus and TMZ
Radiation: WBRT without avoidance of hippocampus — Whole brain radiotherapy of 30Gy/10f by IMRT, with or without boost. The dose of hippocampus is not considered.
  Arms: WBRT; WBRT with TMZ

SUMMARY:
The purpose of this study is to evaluate the effects on neurocognitive function of whole-brain radiotherapy (WBRT) with/without TMZ concurrent chemotherapy or avoidance of hippocampus for patients of brain metastases, as well as the feasibility and risk of avoidance of hippocampus during whole-brain radiotherapy.

DETAILED DESCRIPTION:
This is a phase II randomized clinical trial. It is reported that avoidance of hippocampus during whole-brain radiotherapy (WBRT) had benefits in preservation of memory for patients, and the use of concurrent TMZ in radiotherapy for patients with brain metastases benefited for treating outcome.

The purpose of this study is to evaluate the effects on neurocognitive function of whole-brain radiotherapy with/without TMZ concurrent chemotherapy or avoidance of hippocampus for patients of brain metastases, as well as the feasibility and risk of avoidance of hippocampus during whole-brain radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary lesions diagnosed by pathology or cytology
* Brain metastases confirmed by brain MRI or CT(>3 brain metastases）
* Brain metastases beyond 5mm of hippocampus
* Male or female patients with age between 18 and 75 years old
* Karnofsky Performance Scores ≥ 60
* Expected survival ≥ 6 months
* No previous brain surgery or brain radiotherapy
* Without dysfunction of heart, lung, liver, kidney and hematopoiesis
* The primary carcinoma is under control

Exclusion Criteria:

* MMSE score <27
* Dysfunction of heart, lung, liver, kidney or hematopoiesis
* Severe neurological, mental or endocrine diseases
* History of alcohol or drug abuse within 3 months
* Visual or hearing dysfunction, low education level, or other reasons leading to not capable of taking the MMSE test
* Currently under treatment may effect patients' neurocognitive functions
* Patients participated in clinical trials of other drugs within last 3 months
* Other unsuitable reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of neurocognitive function between baseline and 4 months after radiotherapy | baseline; four months after radiotherapy
  Neurocognitive function is evaluated by Minimum Mental State Examination (MMSE)

SECONDARY OUTCOMES:
Effect on response rate | baseline; One, two, four, six, and twelve months after radiotherapy
  Response is evaluated on basis of RECIST
The tolerance of radiotherapy with TMZ concurrent chemotherapy | baseline; once a week through during radiotherapy, up to 3 weeks
  Adverse effects are evaluated by CTCAE 4.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, Professor, Principal Investigator — Department of Radiation Oncology, Sun Yat-Sen University Cancer Center
Locations (10):
- China (10):
  - Department of Radiation Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Three Nine Brain Hospital, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Guangzhou People's Liberation Army Hospital 421, Guangzhou, Guangdong
  - Panyu Central Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Jinan University, Guangzhou, Guangdong
  - The Affiliated Cancer Hospital Of Guangzhou Medical Collage, Guangzhou, Guangdong
  - Guangdong Provincial Hospital Of Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Guangzhou Medical Collage, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital, Sun Yat-Sen University, Zhuhai, Guangdong